CLINICAL TRIAL: NCT07071168
Title: Developing A Hearing-physical Activity Dual-task Training App for Older Adults With Hearing Loss: A Mixed Method Study
Brief Title: Hearing-physical Activity Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, ZHAO Yan Ivy, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P0054427
Record Dates: First submitted 2025-07-08; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss, Age-Related
MeSH Terms: conditions — Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity group (Experimental): A hearing-physical activity training
  Interventions: Behavioral: hearing-physical activity training
- Control group (Placebo Comparator): waiting list group
  Interventions: Behavioral: hearing-physical activity training

INTERVENTIONS:
Behavioral: hearing-physical activity training — In this study, the intervention was designed to span 10 weeks. Based on our previous study, participants will attend hearing training 30 minutes/day, 5 days/week, The physical activity program will be performed at moderate intensity, 60 min/day, 3 days/week.39

SUMMARY:
Background

By 2050, approximately 2.5 billion people are expected to experience some degree of age-related hearing loss (ARHL). Greater ARHL is associated with decreased communication, reduced physical activity and social engagement, increased depressive symptoms, cognitive decline and a higher risk of dementia. While previous studies highlight the benefits of combing hearing training and physical activity for older adults with ARHL, existing interventions are very limited. Additionally, the development of previous interventions often lacks end-user involvement, resulting in low adherence.

Objectives

This study aims to co-design a hearing-physical activity dual-task training app with older adults with ARHL, the potential end-users; to assess the feasibility and acceptability of the app using based on the theoretical framework of acceptability; and to examine its preliminary effects on improving physical activity, communication, loneliness, depressive symptoms and cognitive functions for older adults with age-related hearing loss.

Hypothesis to be tested

The app is feasible and acceptable to participants. Upon completing the 10-week intervention, the intervention group will report significantly greater improvements in physical activity, communication, loneliness, depressive symptoms and cognitive functions than the control group. These findings will support subsequent investigations in a larger-scale randomized controlled trial.

Research Design and Methods

This study consists of three phases. Phase 1: co-develop a prototype app that combines hearing and physical activity dual-task trainings, incorporating a music therapy component for older adults with ARHL. Co-design workshops will be conducted following the community-based participatory research methodology, where participants will engage in plenary and breakout sessions. Phase 2: conduct a two-arm, single-blinded, pilot randomized controlled trial. Phase 3: conduct individual semi-structured interviews immediately after the intervention. Four process evaluation outcomes will be observed, namely feasibility, fidelity, and acceptability, along with implementation barriers and facilitators. Participants will include Chinese adults aged 60 years or older, with mild-to-moderate HL with a pure-tone average of 20-50 dB across octave frequencies 0.5 to 4kHz in both ears.

Main outcome measures Physical activity levels.

Data analysis

Descriptive statistics, an independent sample t-test or chi square test, generalized estimating equation and thematic analysis will be used.

Expected results

A hearing-physical activity dual-task training app prototype, available in both Cantonese and Mandarin, will be co-designed, tested and refined to a final version. Participants could benefit from incorporating tailored intervention for physical activity with auditory rehabilitation.

ELIGIBILITY:
The inclusion criteria are: (1) ethnic Chinese aged 60 years and above living at home; (2) with mild to moderate hearing loss diagnosed by a pure-tone average of 20 to 50 dB across octave frequencies 0.5 to 4kHz in both ears; and (3) no cognitive impairment [score of ≦2 on the 5-item Abbreviated Memory Inventory for the Chinese (AMIC)].

The exclusion criteria include: (1) those with a diagnosis of a major neurocognitive disorder; (2) a history of symptomatic stroke or other disease of the central nervous system; 3) a serious medical or psychiatric illness (e.g., severe depression, schizophrenia, bi-polar disorder) or a visual impairment that would interfere with using app.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Physical activity | 7 days
  Physical activity levels (objectively): A wrist-worn ActiGraph GT3X+, valid step counter will be used to measure daily step-count. 44 Physical activity levels (subjectively): will be measured using the Chinese version of the 7-item International Physical Activity Questionnaire, which assesses the durations of time in the past 7 days that respondent stayed sedentary or engaged in ambulatory, moderate or vigorous physical activities. It has good psychometrics at the scale- and subscale- levels and significantly correlated with the objective physical activity measures.

SECONDARY OUTCOMES:
Loneliness | 2 weeks
  Loneliness will be measured using the 6-item De Jong Gierveld Loneliness Scale (Chinese version).47 It consists of two subscales: emotional loneliness and social loneliness. The scale has been validated and recommended as reliable (Cronbach's a=0.76, the intra-class correlation coefficients ranged from 0.98 to 1.00).
Communication | 2 weeks
  Communication will be measured using Chinese version of the Hearing Handicap Inventory for the elderly (HHIE)48
Depressive symptoms | 2 weeks
  Depressive symptoms will be measured by PHQ-9, which is a 9-item questionnaire used for screening, diagnosing, monitoring, and measuring the severity of depression
Cognitive function | 2 weeks
  Cognitive function will be measured by the Hong Kong-Montreal Cognitive Assessment (HK-MoCA).

IPD SHARING:
Plan to Share IPD: No